CLINICAL TRIAL: NCT03917732
Title: Randomized Controlled Study to Evaluate the Efficacy of a Cognitive Training Approach to Improve Urinary Dysfunction in Parkinson's Disease
Brief Title: Cognitive Therapy for Urinary Dysfunction in Parkinson´s Disease
Acronym: PD-UD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University of Kiel (Other)
Responsible Party: Principal Investigator, Daniela Berg, Director of the Department of Neurology, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D418/19
Record Dates: First submitted 2019-04-01; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Parkinson Disease; Urinary Disease Other
MeSH Terms: conditions — Parkinson Disease | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive training (Experimental): The cognitive training the investigators are planning consists of three modules which, in their entirety, are intended to help improve bladder dysfunction, which leads to psychological distress in patients: psychoeducation, training of cognitive functions and training in behavioural therapeutic techniques.
  The training will take place over six weeks, with two sessions per week in the first three weeks. In the following three weeks the frequency will be reduced to once a week so that there will be 9 sessions. The duration of each training session is 90 minutes.
  Interventions: Behavioral: cognitive training
- pelvic floor training (Active Comparator): At the beginning of the training, perception of the pelvic floor is the most important factor. The patients should learn the motor skills to consciously perceive and feel the pelvic floor muscles. This requires a lot of concentration and movement control. After this perception phase, the learned movements are internalized. The fine coordination of the pelvic floor muscles is more harmonious and the tensing and relaxing of the muscles becomes easier over time. In the last phase of the training, the movements and muscle activations should be internalised in such a way that they are anchored as automated movement patterns.
  The training will take place over six weeks, with two sessions per week in the first three weeks. In the following three weeks the frequency will be reduced to once a week so that there will be 9 sessions. The duration of each training session is 90 minutes.
  Interventions: Behavioral: pelvic floor training

INTERVENTIONS:
Behavioral: cognitive training — The cognitive training the investigators are planning consists of three modules which, in their entirety, are intended to help improve bladder dysfunction, which leads to psychological distress in patients: psychoeducation, training of cognitive functions and training in behavioural therapeutic techniques.
  The training will take place over six weeks, with two sessions per week in the first three weeks. In the following three weeks the frequency will be reduced to once a week so that there will be 9 sessions. The duration of each training session is 90 minutes.
  Arms: cognitive training
Behavioral: pelvic floor training — At the beginning of the training, perception of the pelvic floor is the most important factor. The patients should learn the motor skills to consciously perceive and feel the pelvic floor muscles. This requires a lot of concentration and movement control. After this perception phase, the learned movements are internalized. The fine coordination of the pelvic floor muscles is more harmonious and the tensing and relaxing of the muscles becomes easier over time. In the last phase of the training, the movements and muscle activations should be internalised in such a way that they are anchored as automated movement patterns.
  The training will take place over six weeks, with two sessions per week in the first three weeks. In the following three weeks the frequency will be reduced to once a week so that there will be 9 sessions. The duration of each training session is 90 minutes.
  Arms: pelvic floor training

SUMMARY:
Idiopathic Parkinson's syndrome (IPS) is one of the most common neurodegenerative diseases. The prevalence and significance of this disease is continuously increasing in the course of demographic change. For many decades, the focus of diagnostics and therapy was on the motor symptoms of IPS. Only in recent years, it has been recognized that Parkinson's patients also suffer from a variety of non-motor symptoms. These have a decisive influence on the patient's quality of life. As one of the most common non-motor symptoms, 55 to 80% of IPS patients suffer from urinary dysfunction. This is associated with a very high impairment of quality of life due to a high degree of stigmatization and impairment of social participation. In clinical everyday life, Parkinson's patients regularly report the occurrence of a strong imperative urge to urinate, which occurs suddenly and is usually triggered by a certain external stimuli. Specific cognitive processing and reflection of these external stimuli seems to help overcome the imperative urge to urinate. From this clinical observation, it can be assumed that the imperative urge to urinate is subject to a certain cognitive control in the sense of targeted inhibition.

The pharmacological therapy of urinary dysfunction in IPS patients is severely restricted and characterized by insufficient proof of efficacy as well as a high potential for side effects. In clinical practice, alpha-blockers and anticholinergics are frequently used, but the evidence base for IPS is inadequate. In addition, there is a highly relevant risk for Parkinson's patients of specific side effects such as orthostatic dysregulation or deterioration of cognition up to psychoses and hallucinations. This greatly limits their use especially in older IPS patients. While the use of dopaminergic medication is essential for the treatment of motor symptoms in Parkinson's patients, a large number of studies have not confirmed sufficient evidence for the efficacy of dopaminergic medication in urinary dysfunction. In addition, non-pharmacological therapy options, in particular pelvic floor training, are used to treat bladder dysfunction. Due to the lack of risk of side effects, pelvic floor training is currently recommended as a first-line therapy option for IPS patients. Initial studies have shown positive effects, but due to the lack of randomized controlled trials, a sufficient evidence base for this has not yet been established.

The aim of the study is to examine whether a purely cognitive therapy approach is suitable to improve subjective and objective symptoms of urinary dysfunction in IPS patients. This therapeutic approach will be compared with the gold standard of pelvic floor training in terms of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* consenting capacity (MOCA >17) and written consent
* idiopathic parkinson syndrome according to UK Brain Bank criteria
* female gender

Exclusion Criteria:

* missing consenting capacity (MOCA <18)
* current depressive episode (BDI > 18)
* current intake of medication for the treatment of bladder dysfunction

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in the International Consultation on Incontinence Questionnaire Overactive Bladder Module (ICIQ-OAB) | 4 weeks before beginning and 4 weeks after completion of the training
  The ICIQ-OAB is a questionnaire for evaluating overactive bladder and related impact on quality of life (QoL) and outcome of treatment in men and women in research and clinical practice across the world. The ICIQ-OAB is derived from the fully validated ICSmale and BFLUTS questionnaires and provides a measure to assess the impact of urinary frequency, urgency, urge incontinence and nocturia symptoms.
Change in the International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol) | 4 weeks before beginning and 4 weeks after completion of the training
  The ICIQ-LUTSqol is a psychometrically robust patient-completed questionnaire evaluating quality of life (QoL) in urinary incontinent patients for use in research and clinical practice across the world. The ICIQ-LUTSqol is the King's Health Questionnaire (KHQ) adapted for use within the ICIQ structure and provides a measure to assess the impact of urinary incontinence on quality of life with particular reference to social effects. It is an ideal research tool as it explores in detail the impact on patients' lives of urinary incontinence and can be used as an outcome measure to assess impact of different treatment modalities.
Change in the Patient Perception of Bladder Condition (PPBC) | 4 weeks before beginning and 4 weeks after completion of the training
  The PPBC is a single-item, global outcome measure for urinary incontinence.
Change in the International Prostate Symptom Score (I-PSS) | 4 weeks before beginning and 4 weeks after completion of the training
  The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
Change in the Uroflowmetric | 4 weeks before beginning and 4 weeks after completion of the training
  Uroflowmetry measures the flow of urine. It tracks how fast urine flows, how much flows out, and how long it takes. It's a diagnostic test to assess how well the urinary tract functions.

SECONDARY OUTCOMES:
Change in the Verbal memory function through the Rey Auditory Verbal Learning Test (RAVLT) | 4 weeks before beginning and 4 weeks after completion of the training
  Participants are given a list of 15 unrelated words repeated over five different trials and are asked to repeat. Another list of 15 unrelated words are given and the client must again repeat the original list of 15 words and then again after 30 minutes.
Change in the Visuomotor abilities and nonverbal memory Rey-Osterrieth complex figure test (ROCF) | 4 weeks before beginning and 4 weeks after completion of the training
  The Rey-Osterrieth complex figure test (ROCF) is a neuropsychological assessment in which patients are asked to reproduce a complicated line drawing, first by copying it freehand (recognition; measures visuomotor abilities), and then drawing from memory (recall; measures nonverbal memory).
Change in the Verbal short term memory functions through the Digit Span test | 4 weeks before beginning and 4 weeks after completion of the training
  Verbal short term memory span measures the number of discrete units over which the patient can successively distribute his attention and still organize them into a working unit. To generalize, it refers to the ability of the patient to reproduce immediately, after one presentation, a series of discrete stimuli in their original order.
Change in the Response inhibition through the Stroop test | 4 weeks before beginning and 4 weeks after completion of the training
  The Stroop test is a widely used measure of selective attention that requires interference resolution, response inhibition, and response selection.
Change in the Visual attention and task switching though the Trial Making Test | 4 weeks before beginning and 4 weeks after completion of the training
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy.
Change in the Word fluency through the Regensburger Word Fluency Test | 4 weeks before beginning and 4 weeks after completion of the training
  In the Regensburger Word Fluency Test patients have to produce as many words as possible from a given category or beginning with a specific letter within 2 minutes.

OTHER OUTCOMES:
Changes in functional magnet resonance imaging (fMRI) within a Go/NoGo paradigm | 4 weeks before beginning and 4 weeks after completion of the training
  The investigators aim to answer the question whether there are different activity patterns in Parkinson's patients with bladder dysfunction compared to Parkinson's patients without bladder dysfunction in the areas involved in bladder function regulation while concerning a Go/NoGo paradigm.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Berg, Prof. Dr., Study Director — Department of Neurology, University Hospital Schleswig- Holstein
Locations (1):
- Department of Neurology, University Hospital Schleswig-Holstein, Kiel, Schleswig-Holstein, Germany